CLINICAL TRIAL: NCT03425305
Title: Serum Uric Acid Levels and Initial Presentation of Cardiovascular Diseases: a CALIBER Study
Brief Title: Serum Uric Acid Levels and Onset of Cardiovascular Diseases: a CALIBER Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: CALIBER 16-176R; RP-PG-0407-10314 (Other Grant/Funding Number: UK National Institute for Health Research); 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2018-01-24; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-11

CONDITIONS: Stable Angina; Unstable Angina; Myocardial Infarction; Unheralded Coronary Heart Disease Death; Heart Failure; Cardiac Arrest; Transient Ischaemic Attack; Ischemic Stroke; Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Peripheral Arterial Disease; Abdominal Aortic Aneurysm; Atrial Fibrillation
Keywords: Serum uric acid; Cardiovascular disease; Atherosclerosis
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Myocardial Infarction; Heart Failure; Heart Arrest; Ischemic Attack, Transient; Ischemic Stroke; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Peripheral Arterial Disease; Aortic Aneurysm, Abdominal; Atrial Fibrillation; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Serum uric acid level is a commonly measured biomarker. The association between serum uric acid level and the risk of developing cardiovascular diseases has been observed in some studies, while others showed controversial results. Estimation of this association may help to predict cardiovascular outcomes and may guide new treatment strategies. The hypothesis is that increased serum uric acid level is associated with a range of cardiovascular diseases.

DETAILED DESCRIPTION:
Smaller observational studies suggested that increased serum uric acid level is associated with increased incidence of several cardiovascular diseases. Associations with specific initial presentations of cardiovascular diseases have not been studied in large cohort from the general population, but may be of interest for use in risk prediction or to guide therapeutic strategies.

The aim of this study is to estimate associations between serum uric acid level and initial presentation of a range of cardiovascular diseases.

The study will use data from the CALIBER dataset of clinically collected electronic health record data from England. Patients enter the study when they have a blood urate measurement recorded in the dataset, and they are followed up until they experience one of the cardiovascular endpoints, death or transfer out of the participating primary care practice.

This study is part of the CALIBER (Clinical disease research using linked bespoke studies and electronic records) programme funded from the National Institute for Health Research (NIHR) and Wellcome Trust. The central theme of the CALIBER research is linkage of the Inpatient Hospital Episode Statistics (HES) with primary care (Clinical Practice Research Datalink) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* Patients registered with a participating general practice during the study period
* Age 30 years or older at study entry
* No record of previous diagnosis of cardiovascular disease
* Follow up for at least one year before the index date.

Exclusion Criteria:

* Patients without a measurement of blood urate level during the study period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort study of patients in the CALIBER database who have a record of a blood urate measurement during the study period while registered at one of 225 general practices contributing data to CPRD (the Clinical Practice Research Datalink) and consenting to data linkage.
Sampling Method: Non-Probability Sample
Enrollment: 180000 (Actual)
Dates: Start 1998-01 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Initial presentation of cardiovascular diseases | 15 years
  First recorded diagnosis of cardiovascular disease during follow-up: Stable angina, unstable angina, myocardial infarction, unheralded coronary heart disease death, heart failure, cardiac arrest/sudden cardiac death, transient ischaemic attack, ischaemic stroke, subarachnoid haemorrhage, intracerebral haemorrhage, peripheral arterial disease, abdominal aortic aneurysm, atrial fibrillation. We will identify the diagnoses using ICD-10 or Read codes in the linked data sources. Definitions for each endpoint are provided on the CALIBER data portal (https://www.caliberresearch.org/portal).

SECONDARY OUTCOMES:
All cause mortality | 15 years

REFERENCES:
- [Background] Denaxas SC, George J, Herrett E, Shah AD, Kalra D, Hingorani AD, Kivimaki M, Timmis AD, Smeeth L, Hemingway H. Data resource profile: cardiovascular disease research using linked bespoke studies and electronic health records (CALIBER). Int J Epidemiol. 2012 Dec;41(6):1625-38. doi: 10.1093/ije/dys188. Epub 2012 Dec 5. PMID 23220717
- [Background] Li X, Meng X, Timofeeva M, Tzoulaki I, Tsilidis KK, Ioannidis JP, Campbell H, Theodoratou E. Serum uric acid levels and multiple health outcomes: umbrella review of evidence from observational studies, randomised controlled trials, and Mendelian randomisation studies. BMJ. 2017 Jun 7;357:j2376. doi: 10.1136/bmj.j2376. PMID 28592419
- [Background] Holme I, Aastveit AH, Hammar N, Jungner I, Walldius G. Uric acid and risk of myocardial infarction, stroke and congestive heart failure in 417,734 men and women in the Apolipoprotein MOrtality RISk study (AMORIS). J Intern Med. 2009 Dec;266(6):558-70. doi: 10.1111/j.1365-2796.2009.02133.x. Epub 2009 May 26. PMID 19563390
- See also: CALIBER web site and data portal — http://www.caliberresearch.org/

DOCUMENTS (1):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03425305/Prot_000.pdf